CLINICAL TRIAL: NCT04829513
Title: Exercise and Two Different Kinesiotape Applications in Addition to Exercise in Patients With Sacroiliac Joint Dysfunction: A Randomized Controlled Study
Brief Title: Exercise and Two Different Kinesiotape Applications in Patients With Sacroiliac Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ufuk University (Other)
Responsible Party: Principal Investigator, Saime Ay, Principal investigator, Ufuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15112016-5
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Sacroiliac Joint Dysfunction

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home Exercise (Active Comparator): The group will be given a home exercise programme involving flexibility and strengthening of the lower back, hip girdle and sacroiliac region.
  Interventions: Procedure: Home Exercise
- Home Exercise and Ligament Correction Kinesiotaping (Active Comparator): In addition to the home exercise program, ligament correction kinesiotaping will be applied to the patients' sacroiliac region.
  Interventions: Procedure: Home Exercise; Procedure: Ligament Correction Kinesiotaping
- Home Exercise and Lymphatic Correction Kinesiotaping (Active Comparator): In addition to the home exercise program, lymphatic correction kinesiotaping will be applied to the patients' sacroiliac region.
  Interventions: Procedure: Home Exercise; Procedure: Lymphatic Correction Kinesiotaping

INTERVENTIONS:
Procedure: Home Exercise — This is a home exercise programme that involves flexibility and strengthening of the waist, hip girdle and sacroiliac region. These exercises are first shown by the physiotherapist in hospital, and then they are asked to do the exercises at home using illustrated forms. Patients continue the exercises as a home programme once a day for 1 month.
Procedure: Ligament Correction Kinesiotaping — Ligament correction kinesiotaping will be applied to the patients' sacroiliac region. Taping will be done once a week. It will be kept for 5 days. This application will be repeated 3 times.
  Arms: Home Exercise and Ligament Correction Kinesiotaping
Procedure: Lymphatic Correction Kinesiotaping — Lymphatic correction kinesiotaping will be applied to the patients' sacroiliac region. Taping will be done once a week. It will be kept for 5 days. This application will be repeated 3 times.
  Arms: Home Exercise and Lymphatic Correction Kinesiotaping

SUMMARY:
This study is a randomized controlled study. 99 patients between the ages of 18-65 who were diagnosed with sacroiliac joint dysfunction will be included in the study.

DETAILED DESCRIPTION:
33 patients will be given a home exercise program that strengthens the waist and hip girdle (to be shown once in the hospital by a physiotherapist and the form of the exercises will be given), 33 patients will be given kinesiotaping (KT) with ligament correction technique with the exercise program, and 33 patients will be given kinesiotaping with lymphatic correction technique with the exercise program. Patients will do the exercises once a day for 1 month. KT will be repeated once a week for 3 weeks. When taping is performed, it will be kept for 5 days.The patients' pain at rest and during movement will be measured using the Visuel Analog Scale (VAS). Patient Global Assessment and Oswestry Disability Index (ODI) will be questioned. Evaluations will be performed before, 4th week and 1 month after treatment (8th week).

ELIGIBILITY:
Inclusion Criteria:

* Patients with sacroiliac joint dysfunction between the ages of 18-65

Exclusion Criteria:

* Patients with rheumatological inflammatory disease
* Inflamatory sacroiliitis
* Patients with polyarthrosis, herniated disc, severe symptomatic disc degeneration, spinal stenosis and spondyloarthrosis.
* Patients with a history of pelvic trauma
* Patients with metabolic bone disease, infection, malignancy, pregnancy
* Patients with open wounds in the lumbar and sacral area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Pain at rest | Before treatment (T1), After treatment at 4th week (T2), Follow-up at 8th week (T3)
  Pain at rest will be measured using the Visuel Analog Scale (0-10 cm).Patients are asked to rate their pain at rest over the past week and to mark a point on a 10 cm line with endpoints '0 = no pain' and '10 = worst pain imaginable'. The distance (cm) measured from the 'no pain' endpoint to the point marked by the patient is reported as the VAS score.
Pain at movement | Before treatment (T1), After treatment at 4th week (T2), Follow-up at 8th week (T3)
  Pain at movement will be measured using the Visuel Analog Scale (0-10 cm).Patients are asked to rate their pain at rest over the past week and to mark a point on a 10 cm line with endpoints '0 = no pain' and '10 = worst pain imaginable'. The distance (cm) measured from the 'no pain' endpoint to the point marked by the patient is reported as the VAS score.

SECONDARY OUTCOMES:
Patient Global Assessment | Before treatment (T1), After treatment at 4th week (T2), Followup at 8th week (T3)
  Patient Global Assessment in the last week will be questioned by Visuel Analog Scale. Patients will be asked to mark their global assessment on a 0-10 cm visual analog scale (0:very good -10: very poor). Lower values indicate better status.
Oswestry Disability Index | Before treatment (T1), After treatment at 4th week (T2), Followup at 8th week (T3)
  Oswestry Disability Index will be questioned to determine the level of disability.The degree of disability is quantified on a scale of 0 to 100%. As the total score increases, the level of disability also increases.

CONTACTS AND LOCATIONS:
Overall Officials: saime ay, Principal Investigator — Ufuk University
Locations (1):
- Ufuk University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No